CLINICAL TRIAL: NCT00414453
Title: Trial of Analgesia With Lidocaine or Extended-release Oxycodone for Neuropathic Pain Treatment in Multiple Sclerosis (TALENT-MS)
Brief Title: Trial of Analgesia With Lidocaine or Extended-release Oxycodone for Neuropathic Pain Treatment in Multiple Sclerosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Did not reach enrollment goals
Sponsor: University of Rochester (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Robert Dworkin, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TALENT-MS
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Results first posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-06

CONDITIONS: Neuropathic Pain; Chronic Pain; Multiple Sclerosis
Keywords: Neuropathic pain; Chronic pain; Multiple sclerosis; Central neuropathic pain; Peripheral neuropathic pain; Opioid analgesic; Lidocaine
MeSH Terms: conditions — Neuralgia; Chronic Pain; Multiple Sclerosis | interventions — Lidoderm; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lidocaine 5% + placebo patch, ER and placebo pills (Active Comparator): 5% lidocaine patch used as intervention placebo patch used with extended release oxycodone or with placebo pills and placebo patches a randomized subjects given extended release oxycodone and placebo patches during this treatment placebo pills used with lidocaine 5% patch group and with placebo patch/placebo pill group period
  Interventions: Drug: Lidocaine patch 5%; Drug: Extended-release oxycodone; Drug: Placebo extended-release oxycodone pills; Drug: Placebo lidocaine patches

INTERVENTIONS:
Drug: Lidocaine patch 5% — lidocaine 5% patch; 12 hours on, 12 hours off
  Other Names: Lidoderm
Drug: Extended-release oxycodone — extended-release oxycodone titrating schedule
  Other Names: Oxycontin
Drug: Placebo extended-release oxycodone pills — placebo pills with titrating schedule
  Other Names: Placebo pill
Drug: Placebo lidocaine patches — used with extended release oxycodone group; used with placebo pills/placebo patches
  Other Names: Placebo patch

SUMMARY:
This study will determine whether treatment with an extended-release opioid or topical lidocaine is effective in relieving distal symmetric lower extremity burning pain associated with multiple sclerosis (MS). If treatment with topical lidocaine is efficacious, it will have important implications for understanding this chronic pain syndrome, which is widely assumed to be caused by central nervous system pathology.

DETAILED DESCRIPTION:
This study is a single-center, double-blind, 15-week, 3-period crossover clinical trial. Subjects will complete each of the following 5-week long periods (unless they withdraw from the trial): 1) placebo pills and topical lidocaine patches, 2)extended-release oxycodone pills and placebo(vehicle) patches, and 3)placebo pills and placebo patches. Sixty subjects will be randomized to one of 6 treatment sequences. It is expected that this trial will take approximately 2 years to complete.

ELIGIBILITY:
Inclusion Criteria:

* "Definite MS" as defined by revised McDonald criteria.
* Bilateral distal symmetric burning pain involving both feet for at least three months.
* Baseline weekly average pain rating equal to four or greater on 0-10 numerical scale.
* Stable MS medication and pain-related medications for 8 weeks prior to screening.
* Must come to Research Center for appointments

Exclusion Criteria:

* Topical treatment with lidocaine, capsaicin, or other topical analgesics within 3 months prior to screening.
* Any treatment with opioid analgesics or tramadol within 3 months prior to screening.
* Hypersensitivity to Lidoderm, lidocaine, or other local anesthetics.
* Hypersensitivity or inability to tolerate opioid analgesics.
* Current treatment with a total of 3 or more antidepressant or anticonvulsant drugs for pain.
* Current treatment with Class I anti-arrhythmic agents at baseline.
* Beck Depression Inventory score > 16 or clinically significant depression or dementia.
* History of suicide attempt or current intent or plan.
* History of excessive alcohol use or any illicit drug use within the past 2 years.
* Lack of adequate birth control in pre-menopausal women of childbearing age.
* Other pain more severe than lower extremity burning pain.
* Open skin lesions in the area where the lidocaine patch is to be applied.
* Cancer within the previous 5 years other than skin cancer.
* MS exacerbation or any treatment with corticosteroids within 3 months prior to screening.
* History of peripheral neuropathy, lower limb amputation, or another neuromuscular syndrome or systemic disorder known to be associated with sensory neuropathy.
* Does not meet criteria of baseline lab values at screening visit.
* Nerve conduction studies consistent with peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Dworkin, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7-6-2006 to 9-23-2008 at the medical center
Pre-assignment Details: 19 subjects were enrolled in this study however the study was terminated due to not reaching enrollment goals in a timely manner. Therefore there was no data analysis completed for this study. We do not have randomization data for these participants because the data is not available and is locked.
Groups:
- Lidocaine 5% + Placebo Patch, ER + Placebo Pills: 5% lidocaine patch used as intervention Lidocaine patch 5%: lidocaine 5% patch; 12 hours on, 12 hours off
  placebo patch used with extended release oxycodone or with placebo pills and placebo patches arm Placebo lidocaine patches: used with extended release oxycodone group; used with placebo prandomized subjects given extended release oxycodone and placebo patches during this treatment period
  Extended-release oxycodone: extended-release oxycodone titrating scheduleills/placebo patches
  placebo pills used with lidocaine 5% patch group and with placebo patch/placebo pill group
  Placebo extended-release oxycodone pills: placebo pills with titrating schedule
Period: Overall Study
Arm/Group | Lidocaine 5% + Placebo Patch, ER + Placebo Pills
Started | 19
Completed | 3
Not Completed | 16
Not completed — Abnormal lab work | 16

BASELINE CHARACTERISTICS:
Arm/Group | Lidocaine 5% + Placebo Patch, ER + Placebo Pills
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Diary Pain Ratings During Final Week of Each Treatment Period
Description: subject identifies daily pain rating during final week of each treatment period using a numeric rating scale
Time Frame: Daily
Population: Data was not analyzed because we the data is locked and is not available.
Groups:
- Lidocaine Patch 5%: 5% lidocaine patch used as intervention
  Lidocaine patch 5%: lidocaine 5% patch; 12 hours on, 12 hours off
- Placebo Patch: placebo patch used with extended release oxycodone or with placebo pills and placebo patches arm
  Placebo lidocaine patches: used with extended release oxycodone group; used with placebo pills/placebo patches
- Extended Release Oxycodone: randomized subjects given extended release oxycodone and placebo patches during this treatment period
  Extended-release oxycodone: extended-release oxycodone titrating schedule
- Placebo Pills: placebo pills used with lidocaine 5% patch group and with placebo patch/placebo pill group
  Placebo extended-release oxycodone pills: placebo pills with titrating schedule
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Tolerability (e.g., Number of Adverse Effects, Number of Drop-outs)
Description: subject is questioned regarding any adverse events that have occured since the last contact; also subject can document any issues on daily pain rating diaries
Time Frame: rating of adverse events occur at each visit
Population: Data was not analyzed because we did not reach our enrollment goal and the study was terminated. Data was not analyzed because we the data is locked and is not available.
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Safety (i.e., Number of Serious Adverse Events)
Description: Subject is asked about any adverse events that may have occurred since last contact; also subject can document any adverse events on daily pain diary scales
Time Frame: rating and review of any adverse events occurs at each visit
Population: as for outcome 2
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Brief Pain Inventory Interference Items
Description: subject completes the brief pain questionaire
Time Frame: occurs Visit 1, 3,4,5
Population: as for outcome 2
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Daily Diary Sleep Interference Ratings
Description: Subject identifies degree of sleep interference on a daily basis
Time Frame: daily
Population: Data was not analyzed because we did not reach our enrollment goal and the study was terminated.. Data was not analyzed because we the data is locked and is not available.
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Beck Depression Inventory
Description: Subject completes Beck questionaire
Time Frame: occurs at Visit 1, 3, 4 and 5
Population: as for outcome 2
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Short-form Health Survey 36 (SF-36)
Description: Subject completes short form health survey 36 questionaire
Time Frame: Occurs at Visit 1, 3, 4 and 5
Population: as for outcome 2
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Short-Form McGill Pain Questionnaire
Description: Subject completes short form McGill Pain questionaire
Time Frame: Occurs Visit 1, 3, 4 and 5
Population: as for outcome 2
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Patient Global Impression of Change Scale
Description: Subject completes patient global impression questionaire of change scale
Time Frame: Occurs Visit 3, 4, 5
Population: as for outcome 2
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Kurtzke Expanded Disability Status Scale
Description: Subject completes questionaire on functional status
Time Frame: Occurs at Visit 1
Population: as for outcome 2
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were not collected.
Arm/Group | Lidocaine Patch 5% | Placebo Patch | Extended Release Oxycodone | Placebo Pills
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No